CLINICAL TRIAL: NCT01688050
Title: TRANSFIX - Zenith® TX2® Low Profile Endovascular Graft for Blunt Thoracic Aortic Injury
Brief Title: TRANSFIX Zenith® Transection Clinical Study
Acronym: TRANSFIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-004
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Results first posted 2015-11-18 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Thoracic Aorta; Thoracic Injuries; Blunt Injuries
Keywords: Blunt thoracic aortic injury; Transection; Endovascular graft
MeSH Terms: conditions — Thoracic Injuries; Wounds, Nonpenetrating

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Endovascular Repair (Experimental)
  Interventions: Device: Zenith® TX2® Low Profile Endovascular Graft

INTERVENTIONS:
Device: Zenith® TX2® Low Profile Endovascular Graft — Treatment of Blunt thoracic aortic injuries (BTAIs)
  Other Names: Zenith Alpha Thoracic™ Endovascular Graft

SUMMARY:
The TRANSFIX study is a clinical trial approved by US FDA to study the safety and effectiveness of the Zenith® TX2® Low Profile Endovascular Graft for treatment of Blunt Thoracic Aortic Injury.

ELIGIBILITY:
Inclusion Criteria:

* Vessels suitable for endovascular access and stent graft placement
* Blunt thoracic aortic injury of the descending thoracic aorta
* At least 16 years of age
* Informed consent given by patient or legally authorized representative

Exclusion Criteria:

* Clinical considerations that would compromise patient safety or study outcomes
* Unsuitable arterial anatomy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01-23 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2019-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Starnes, MD, Principal Investigator — University of Washington - Harborview, Division of Vascular Surgery
Locations (21):
- United States (21):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Keck Hospital of USC, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Miami School of Medicine, Miami, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers University, Newark, New Jersey
  - University of North Carolina Vascular Surgery, Chapel Hill, North Carolina
  - University of Cincinnati University Hospital, Cincinnati, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee Medical School, Knoxville, Tennessee
  - UT Southwestern Medical Center - Parkland Memorial Hospital, Dallas, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - University of Washington - Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Starnes BW, Dwivedi A, Giglia J, Woo K, Yeh C; TRANSFIX Study Investigators. Updated outcomes from the TRANSFIX study to evaluate endovascular repair of blunt thoracic aortic injuries with the Zenith Alpha thoracic device. J Vasc Surg. 2020 Jun;71(6):1851-1857. doi: 10.1016/j.jvs.2019.05.070. Epub 2020 Feb 1. PMID 32014287
- [Derived] Starnes BW, Dwivedi AJ, Giglia JS, Woo K, Yeh C; TRANSFIX Study Investigators. Endovascular repair for blunt thoracic aortic injury using the Zenith Alpha low-profile device. J Vasc Surg. 2015 Dec;62(6):1495-503.e1. doi: 10.1016/j.jvs.2015.07.098. Epub 2015 Sep 26. PMID 26391458

RESULTS

PARTICIPANT FLOW:
Groups:
- Endovascular Repair: Zenith® TX2® Low Profile Endovascular Graft
Period: Overall Study
Arm/Group | Endovascular Repair
Started | 50
5-Year | 22 (Patients eligible for Follow-up at 5 year)
Completed | 19
Not Completed | 31
Not completed — Death | 7
Not completed — Conversion to open repair | 1
Not completed — Lost to Follow-up | 13
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 44

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Time Frame: 30 days
Population: One death was adjudicated as unrelated by the Clinical Events Committee (CEC).
Measure: Number; unit: participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 50
participants | 1
Statistical Analysis 1: Comparison: Endovascular Repair; Test type: Other — The primary safety endpoint of this study is analyzed using only descriptive statistics and it is not analyzed for the purpose of statistical inference; All-cause mortality rate (%) = 2.0, 95% CI 2-sided [0 to 5.88] — Wald method

2. Primary Outcome: Aortic Injury-related Mortality
Description: Any death determined by the independent clinical events committee to be causally related to the initial implant procedure, secondary intervention, or rupture of the transected aorta.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 50
participants | 0
Statistical Analysis 1: Comparison: Endovascular Repair; Test type: Other — [test comment as in outcome 1, analysis 1]; Aortic injury-related mortality rate (%) = 0, 95% CI 2-sided [0 to 7.1] — Exact method

3. Primary Outcome: Device Success
Description: Technical success (successful access, deployment, and patency of the Zenith® TX2® Low Profile Endovascular Graft), and freedom from the following: device collapse, type I or type III endoleaks requiring reintervention, and conversion to open surgical repair.
Time Frame: 30 days
Population: One patient had device compression (counted as a failure conservatively although the compression was not consistent with collapse of the proximal end of the device) and one patient had a site-reported Type I endoleak requiring secondary intervention.
Measure: Number; unit: participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 50
participants | 48
Statistical Analysis 1: Comparison: Endovascular Repair; Test type: Other — The primary effectiveness endpoint of this study is analyzed using only descriptive statistics and it is not analyzed for the purpose of statistical inference; Device success rate (%) = 96.0, 95% CI 2-sided [90.6 to 100] — Wald method

ADVERSE EVENTS:
Time Frame: 5-Year
Arm/Group | Endovascular Repair
All-Cause Mortality (participants affected / at risk) | 7/50
Serious Adverse Events (participants affected / at risk) | 30/50
Other Adverse Events (participants affected / at risk) | 21/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular Repair (N=50)
Anaemia (Blood and lymphatic system disorders) | 2 (3)
Arrhythmia (Cardiac disorders) | 3 (3)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Aorto-oesophageal fistula (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Multiple organ dysfunction (General disorders) | 3 (3)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 9 (10)
Urinary Tract Infection (Infections and infestations) | 2 (3)
Abscess limb (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
CNS ventriculitis (Infections and infestations) | 1 (1)
Groin infection (Infections and infestations) | 1 (1)
Pancreatic abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (3)
Tooth abscess (Infections and infestations) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) — Right Labral tear s/p fall down 3-4 stairs while carrying boxes/moving 07-01-2016 Right hip replacement 7-10-2016
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (2)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 4 (5)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) — One additional stroke event was reported. However, per evaluation by the site, the event was not considered to be a serious adverse event. Therefore, it is not present in this table
Carotid artery dissection (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Quadriplegia (Nervous system disorders) | 1 (1)
Device failure (Product Issues) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Haemothroax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Hip Disarticulation (Surgical and medical procedures) | 1 (1) — Extremity left hip disarticulation wound infection: infected hematoma and necrotic muscle
Hip arthroplasty (Surgical and medical procedures) | 1 (1) — orthopaedic surgery (hip replacement and plate removal from tibia)
Withdrawal of life support (Surgical and medical procedures) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) — Hypotension secondary to nausea/vomiting and dehydration
Vascular access site complication (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular Repair (N=50)
Arrhythmia (Cardiac disorders) | 4 (4)
Pneumonia (Infections and infestations) | 8 (8)
Urinary tract infection (Infections and infestations) | 5 (7)
Deep vein thrombosis (Vascular disorders) | 4 (5)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Vascular stent thrombosis (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-06-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT01688050/Prot_SAP_000.pdf